CLINICAL TRIAL: NCT04462874
Title: Mean Systemic Filling Pressure Trends in Liver Transplant Recipients - a Prospective Observational Pilot Trial
Brief Title: Mean Systemic Filling Pressure Trends in Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS - Liver Transplant-4
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-09

CONDITIONS: Liver Transplant; Complications; Liver Diseases; Hemodynamic Instability
Keywords: liver transplantation; mean systemic filling pressure; advanced hemodynamic monitoring; liver cirrhosis
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with end stage liver disease undergoing liver transplantation have varying degrees of intraoperative haemodynamic unstability during various phases of transplantation. It is difficult to determine the cause for hemodynamic instability in these patients and to predict the best treatments. Currently, cardiovascular resuscitation options are triggered by arterial pressure and cardiac output (CO) measures, focusing on the oxygen delivery side of the circulation. The primary determinants of cardiac output reside on the venous side. Veins are 30-50 times more compliant than arteries and contain approximately 75% of the total blood volume. Mean systemic filling pressure provides vital information on this venous side of the circulation. Mean systemic filling pressure , which is defined as the pressure equal to the pressure which would be measured if the heart should suddenly stop pumping and all (arterial and venous) the pressures in the entire circulatory system should be brought to equilibrium instantaneously, is a good, complete and reliable reflection of the total intravascular fluid compartment. We would study the Mean systemic filling pressure in liver transplant recipients and record hemodynamic, respiratory, cardiac and renal function prospectively. Follow up data for 7 days for respiratory, cardiac and renal complications will be collected, along with hospital stay, ICU stay and mortality. The association between Mean systemic filling pressure and these outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing liver transplantation 18-65 years

Exclusion Criteria:

* pregnant patients acute liver failure, acute on chronic liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with liver diseases undergoing liver transplantation
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
mean systemic filling pressures(MSFP) | 1 day
  MSFP trends during liver transplantation, hourly

SECONDARY OUTCOMES:
icu stay | 28 days
  duration of stay in the intensive care unit
28 day mortality | 28 days
  mortality by all causes till day 28

OTHER OUTCOMES:
respiratory complications | 7 days
  number of participants needing reintubation, prolonged mechanical ventilation, intercostal drain placement
acute kidney injury(AKI) | 7 days
  AKI incidence upto 7 days
cardiac complication | 7 days
  number of participants with significant arrhythmias and ischemia associated with hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Karthik T Ponnappan, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India